CLINICAL TRIAL: NCT00723905
Title: Remicade Infusion Management Program
Acronym: RemiTRAC
Status: Completed | Type: Observational
Sponsor: Janssen Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR100746; P04466 (Other: Janssen Inc.)
Record Dates: First submitted 2008-07-25; First posted 2008-07-29 (Estimated); Last update posted 2013-01-15 (Estimated); Status verified 2013-01

CONDITIONS: Crohn Disease; Arthritis, Rheumatoid
Keywords: Crohn's Disease, Rheumatoid Arthritis
MeSH Terms: conditions — Crohn Disease; Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Janssen Inc. plans to collect data on about 3000 to 5000 infliximab infusions per year, starting in the third quarter of 2005. It is expected that about 12 sites from the Remicade Infusion Network (R.I.N.) will participate. This registry will be a multicentre, prospective, observational program that will gather and analyze data on subjects being treated with infliximab.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a good candidate to receive infliximab as per the Product Monograph
* Subject is prescribed infliximab by an appropriate physician
* Subject receives infusion in a community infusion centre.
* Subject has signed the approved consent form.

Exclusion Criteria:

* Not specified in the protocol

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The data captured and reported in this registry will reflect a "real world" approach to the treatment of Rheumatoid Arthritis and Crohn's Disease with infliximab.
Sampling Method: Non-Probability Sample
Enrollment: 1630 (Actual)
Dates: Start 2005-08; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Type and frequency of infusion reactions | Up to 7 years
Pre-infusion treatments and efficacy | Up to 7 years
Infusion reaction management approaches | Up to 7 years
The number of subjects with adverse events | Up to 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Inc. Clinical Trial, Study Director — Janssen Inc.
Locations (2):
- Canada (2):
  - Montreal, Quebec
  - Pointe-Claire

REFERENCES:
- [Derived] Choquette D, Faraawi R, Chow A, Rodrigues J, Bensen WJ, Nantel F. Incidence and Management of Infusion Reactions to Infliximab in a Prospective Real-world Community Registry. J Rheumatol. 2015 Jul;42(7):1105-11. doi: 10.3899/jrheum.140538. Epub 2015 Jun 15. PMID 26077415